CLINICAL TRIAL: NCT06784596
Title: The Effect of Tele-Consultation Supported Education Based on Watson's Theory of Human Caring on Daily Living Activities, Quality of Life, and Self-Care Ability in Patients Undergoing Total Knee Arthroplasty
Brief Title: The Effect of Tele-Consultation Supported Education After Total Knee Arthroplasty Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turgut Sohret (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Sponsor-Investigator, Turgut Sohret, Researcher, Ataturk Training and Research Hospital
Organization: Ataturk Training and Research Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ATATURKTRH-Nursing-TS-02
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Knee Arthroplasty, Total
Keywords: total knee replacement; education; teleconsulting; activities of daily living; self-care ability; quality of life

STUDY DESIGN:
Intervention Model Description: A design with two groups, one experimental and one control group
Who Masked: Participant
Masking Description: Patients were not told which group they were in. In this way, single blinding was achieved.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group provided with teleconsulting supported training (Experimental): This group will be the group that will receive training and teleconsultancy services.
  Interventions: Other: Teleconsulting supported training
- Group provided with standard care (No Intervention): This group will only be monitored with standard care and will not receive education or telecounseling.

INTERVENTIONS:
Other: Teleconsulting supported training — Patients in this group will be provided with training the day before surgery, on the morning of surgery and on the day of discharge, and will receive teleconsulting services at the 1st, 2nd, 3rd, 4th, 5th, 6th, 8th, 10th and 12th weeks after discharge. will be given.
  Arms: Group provided with teleconsulting supported training

SUMMARY:
Following total knee arthroplasty, patients may encounter numerous problems that can hinder the performance of daily living activities, negatively impact quality of life, and increase morbidity and mortality rates. In this context, this study was designed to evaluate the effect of nursing education and tele-consultation, based on Watson's Theory of Human Caring, on daily living activities, self-care agency, and quality of life in patients undergoing total knee arthroplasty.

DETAILED DESCRIPTION:
Type of the Study This research was designed as a quasi-experimental study with a pre-test and post-test control group. Initially, data will be collected from the "control group" patients receiving routine care. Subsequently, data will be gathered from the "intervention group" patients who will receive an education program supported by tele-consultation and based on Watson's Theory of Human Caring.

Study Location and Timeframe This study will be conducted in the Orthopedics Clinic of Van Yüzüncü Yıl University Research Hospital between March 2025 and March 2026.

Study Population and Sample The study population will consist of patients undergoing total knee arthroplasty at the Orthopedics Clinic of Van Yüzüncü Yıl University Research Hospital , affiliated with the University of Health Sciences, between March 2025 and March 2026. The sample will include patients who agree to participate and meet the inclusion criteria. A power analysis was conducted to determine the sample size using G*Power 3.1 software. Based on a similar study by Bozdemir and Aygin (2021), the effect size was determined as 0.632. To ensure a study power of over 95% at a 5% significance level and with an effect size of 0.632, a minimum of n=55 participants per group was required. Considering a potential 10% loss due to disease and treatment-related factors, it was planned to work with a total of 122 patients.

Variables of the Study Dependent Variables: Average scores of daily living activities, quality of life, and self-care agency

* Independent Variables: Education and tele-consultation based on Watson's Theory of Human Caring
* Control Variables: Patient age, marital status, gender, surgical history, education level, and comorbid conditions

Data Collection Tools

The following tools will be used to collect the research data:

* Patient Identification Form
* KATZ Activities of Daily Living Scale
* Lawton Brody Instrumental Activities of Daily Living Scale
* SF-36 Quality of Life Scale
* Self-Care Agency Scale
* Telephone Follow-up Assessment Form

Patient Identification Form This form was developed by the researchers based on literature to collect demographic data. It includes 12 questions regarding age, gender, phone number, marital status, number of children, educational level, occupation, income status, smoking and alcohol consumption, chronic illnesses, and previous surgical experiences.

KATZ Activities of Daily Living Scale This scale is used to assess basic activities of daily living. It evaluates the level of dependence in six fundamental self-care activities: bathing, dressing, toileting, mobility, continence, and feeding. The total score range is 0-6, where lower scores indicate higher dependence. The scale classifies as dependent (0-2 points), semi-dependent (3-4 points), and independent (5-6 points).

Lawton Brody Instrumental Activities of Daily Living Scale This scale was developed to evaluate instrumental activities in daily life. It consists of eight items, including using a telephone, shopping, preparing meals, housekeeping, laundry, transportation, managing medications, and handling finances. The total score range is 0-8, with lower scores indicating higher dependence.

SF-36 Quality of Life Scale SF-36 is one of the most widely used tools to assess quality of life. It allows users to self-evaluate, can be filled out in a short time, and provides a highly sensitive measurement. The SF-36 examines eight subdimensions of health (physical functioning, physical role, emotional role, pain, mental health, vitality, social functioning, and general health perception) and contains 36 questions. The second question asks about changes in the past year, while the other questions focus on the last four weeks. The fourth and fifth questions are in yes/no format, while the remaining questions use Likert-type scales (3, 5, and 6 points). Additionally, some questions are reverse-coded, and the scores are adjusted accordingly. The total score for each subscale ranges from 0 to 100, with an increase indicating better quality of life and a decrease indicating poorer quality of life.

Self-Care Agency Scale This scale was created to evaluate individuals' ability to perform self-care. The scale assesses four main aspects: "active or passive response to situations," "motivation," "knowledge of health practices," and "self-worth." The scale is answered using a 5-point Likert scale (0: Doesn't describe me at all, 1: Doesn't describe me very well, 2: I have no idea, 3: Describes me a little, 4: Describes me very well). In the Turkish version, 28 items (such as items 3, 6, 9, 13, 19, 22, 26, 31) are scored negatively and the scoring is done in reverse. Higher scores indicate greater ability and strength in self-care.

Telephone Follow-up Assessment Form This form is designed to evaluate the attitude of the tele-consultation provider, the sufficiency of the information provided, and overall satisfaction with the telephone consultation. The assessment form consists of 7 questions.

Application of Data Collection Tools After obtaining the necessary permissions, the study will include patients who agree to participate and meet the inclusion criteria between March 2025 and March2026 at the Orthopedic Clinic of the Van Yüzüncü Yıl University Research Hospital.

Patients undergoing Total Knee Prosthesis (TKP) surgery will come to the hospital one day before the surgery to complete pre-operative preparations. Depending on the patient's general condition, they will be discharged after at least 2 days of hospitalization. Data will be collected through face-to-face interviews on the day the patients are admitted for surgery, on the day of surgery, and on the day of discharge. Subsequent data will be collected via telephone after the educational program supported by tele-consultation at the 3rd, 6th, and 12th weeks.

Before beginning the data collection, the study's purpose will be explained to the patients undergoing Total Knee Prosthesis (TKP) surgery, and informed consent will be obtained. After obtaining both verbal and written consent, the scale forms will be collected by the researcher.

For the intervention group:

* Pre-Surgery Day: The researcher will visit the patient, explain the purpose of the study, and obtain verbal and written consent. The following scales will be administered: "Patient Identification Form," "KATZ Activities of Daily Living Scale," "Lawton Brody Instrumental Activities of Daily Living Scale," "SF-36 Quality of Life Scale," and "Self-Care Agency Scale."
* Post-Surgery Day: Before the surgery, the "KATZ Activities of Daily Living Scale," "Lawton Brody Instrumental Activities of Daily Living Scale," "SF-36 Quality of Life Scale," and "Self-Care Agency Scale" will be applied.
* Post-Discharge: Before discharge, the same scales will be applied. Then, patients will receive discharge education based on the human care theory.
* Post-Discharge Follow-up: Following the ERAS protocol, patients will be contacted within 24-48 hours after discharge to assess their condition via telephone. Additionally, follow-up consultations will be conducted weekly during the 1st, 2nd, 3rd, 4th, 5th, 6th, 8th, 10th, and 12th weeks via video call on WhatsApp, offering tele-consultation services. At the end of the 3rd, 6th, and 12th weeks, the same scales will be administered again via telephone after tele-consultation.

For the control group:

* Pre-Surgery Day: The researcher will meet with the patient, explain the purpose of the study, and obtain verbal and written consent. The following scales will be administered: "Patient Identification Form," "KATZ Activities of Daily Living Scale," "Lawton Brody Instrumental Activities of Daily Living Scale," "SF-36 Quality of Life Scale," and "Self-Care Agency Scale."
* Surgery Day: Before the surgery, the same scales will be applied.
* Post-Surgery Day: Before discharge, the same scales will be administered face-to-face.
* Post-Discharge Follow-up: At the 3rd, 6th, and 12th weeks, the scales will be collected via telephone. No additional interventions will be given beyond standard care for the control group.

Preparation of the Training Manual The training and training manual will utilize the core concepts of the Human Care Theory, including interpersonal care relationships, care moments, care situations, and healing processes. To ensure that the perioperative process sequence remains intact and to facilitate better understanding for the patient, the manual will be organized under headings such as information on the knee joint, osteoarthritis, total knee prosthesis, preoperative period, intraoperative period, postoperative period, and discharge period.

The prepared training manual will be sent for expert review and, if deemed appropriate, will be applied to the patients. During both the preoperative and pre-discharge education, a training environment will be created based on the Human Care Theory.

The preoperative education and education provided before discharge are expected to last 45-60 minutes. Immediately after the education given on the day before surgery, the training manual will be introduced and handed over to the patient.

Teleconsultation Implementation Guide The goal of the teleconsultation service is to monitor patients following total knee prosthesis surgery, address issues related to the specific educational topics post-surgery, identify problems experienced by the patient, and plan solutions. The teleconsultation service will be offered during the 1st, 2nd, 3rd, 4th, 5th, 6th, 8th, 10th, and 12th weeks. The consultation protocol, developed by the researcher using the core concepts of the Human Care Theory-such as interpersonal care relationships, care moments and situations, and healing processes-will be applied to address the patient's consultation needs.

Consultations will be conducted via video calls, with each session expected to last approximately 30 minutes. If necessary, this duration may be extended. The date and time for each consultation will be arranged with the patient via video call. After each consultation, the timing for the next session will be determined based on the patient's availability. Prior to each consultation, a review of the previous week's topics will be conducted with the patient. Positive feedback will be provided regarding what the patient did correctly, while any mistakes will be addressed with accurate information.

Additionally, reminder messages will be sent to the patient three times a day, based on the contents of the consultation protocol. The researcher, Turgut ŞÖHRET's phone number will be shared with the patient, and the patient will be informed that they may call at any time if needed.

Following the consultations during the 3rd, 6th, and 12th weeks, the following scales will be administered to the patient:

* KATZ Activities of Daily Living Scale
* Lawton Brody Instrumental Activities of Daily Living Scale
* SF-36 Quality of Life Scale
* Self-Care Power Scale

Data Evaluation The data will be collected by PhD student Turgut ŞÖHRET. Statistical analysis and processing of the data will be conducted using the Statistical Package for the Social Sciences (SPSS). The data analysis will be carried out by a statistics expert. Once the data is ensured to be blinded, coded, and labeled, it will be sent to the statistician for analysis. The data will be analyzed using SPSS for Windows version 22. Statistical significance will be considered at a p-value of 0.05, with a Type 1 error rate of 5%, and a 95% confidence interval will be used for evaluation. The normality distribution of the data will be determined by Kurtosis and Skewness coefficients (±2). For the analysis, numbers, percentages, means, and standard deviations will be calculated. For comparisons of binary groups, the independent samples t-test will be used for measurements showing normal distribution, while the Mann-Whitney U test will be used for measurements that do not show normal distribution. For within-group comparisons of binary groups, the paired samples t-test will be used for normally distributed measurements, and the Wilcoxon test will be used for measurements that do not follow normal distribution.

Ethical Principles of the Research Ethical approval for the research has been obtained from the Atatürk University Faculty of Medicine Ethics Committee. Necessary legal permissions will be obtained from Van Yüzüncü Yıl University Research Hospital for conducting the study. The voluntary participation of individuals in the study is of paramount importance, as per the information provided to all participants. After explaining the purpose of the study and how the findings will be used, oral consent will be obtained from the participants (informed consent principle). The principle of "Respect for Autonomy" will be adhered to by ensuring that participants are free to decide whether or not to participate in the study. Participants' information will remain confidential, in line with the principle of "Confidentiality and Protection of Privacy." Throughout the study, individual rights will be protected, and respect for human rights will be ensured, in accordance with the Declaration of Helsinki.

Limitations and Strengths of the Study Since the study will be conducted at Van Yüzüncü Yıl University Research Hospital, the results of the research can only be generalized to patients with characteristics similar to those in the sample group. Additionally, the teleconsultation service will be conducted via video calls, and the possibility that some patients may not own a smartphone is a limitation of the study.

The strengths of the study include the use of a randomized controlled design, the long-term follow-up of patients for three months, and the application of the Human Care Theory, which places significant emphasis on care, making this a strong aspect of the research.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who voluntarily consent to participate,
* Aged 18 years or older,
* Those scheduled for their first Total Knee Arthroplasty (TKA),
* Patients undergoing unilateral knee prosthesis surgery,
* Patients without verbal communication barriers for face-to-face and telephone interactions,
* Patients who own a smartphone and have the WhatsApp application installed.

Exclusion Criteria:

* Patients undergoing Total Knee Arthroplasty (TKA) as an emergency surgical intervention,
* Patients diagnosed with any psychiatric disorder,
* Patients who wish to withdraw from the study voluntarily,
* Patients whose communication is interrupted before the completion of the data collection phase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
KATZ Activities of Daily Living Scale | 1 day
  The scale was developed in 1963 by Katz and his colleagues to assess individuals' basic activities of daily living. This scale measures the level of dependency in six basic self-care activities: bathing, dressing, toileting, transferring, continence, and feeding. The total score ranges from 0 to 6, with lower scores indicating a higher level of dependence. The scale classifies as follows: 0-2 points indicates dependent, 3-4 points indicates partially dependent, and 5-6 points indicates independent.
KATZ Activities of Daily Living Scale | 2 day
  The scale was developed in 1963 by Katz and his colleagues to assess individuals' basic activities of daily living. This scale measures the level of dependency in six basic self-care activities: bathing, dressing, toileting, transferring, continence, and feeding. The total score ranges from 0 to 6, with lower scores indicating a higher level of dependence. The scale classifies as follows: 0-2 points indicates dependent, 3-4 points indicates partially dependent, and 5-6 points indicates independent.
KATZ Activities of Daily Living Scale | 3 weeks
  The scale was developed in 1963 by Katz and his colleagues to assess individuals' basic activities of daily living. This scale measures the level of dependency in six basic self-care activities: bathing, dressing, toileting, transferring, continence, and feeding. The total score ranges from 0 to 6, with lower scores indicating a higher level of dependence. The scale classifies as follows: 0-2 points indicates dependent, 3-4 points indicates partially dependent, and 5-6 points indicates independent.
KATZ Activities of Daily Living Scale | 6 weeks
  The scale was developed in 1963 by Katz and his colleagues to assess individuals' basic activities of daily living. This scale measures the level of dependency in six basic self-care activities: bathing, dressing, toileting, transferring, continence, and feeding. The total score ranges from 0 to 6, with lower scores indicating a higher level of dependence. The scale classifies as follows: 0-2 points indicates dependent, 3-4 points indicates partially dependent, and 5-6 points indicates independent.
KATZ Activities of Daily Living Scale | 12 weeks
  The scale was developed in 1963 by Katz and his colleagues to assess individuals' basic activities of daily living. This scale measures the level of dependency in six basic self-care activities: bathing, dressing, toileting, transferring, continence, and feeding. The total score ranges from 0 to 6, with lower scores indicating a higher level of dependence. The scale classifies as follows: 0-2 points indicates dependent, 3-4 points indicates partially dependent, and 5-6 points indicates independent.
Lawton Brody Activities of Daily Living Scale | 1 day
  The scale was developed in 1969 by Lawton and Brody to assess individuals' instrumental activities of daily living. This scale includes a total of eight items: using the telephone, shopping, preparing meals, housekeeping, doing laundry, traveling, managing medications, and handling finances. The total score ranges from 0 to 8, with lower scores indicating a higher level of dependence.
Lawton Brody Activities of Daily Living Scale | 2 day
  The scale was developed in 1969 by Lawton and Brody to assess individuals' instrumental activities of daily living. This scale includes a total of eight items: using the telephone, shopping, preparing meals, housekeeping, doing laundry, traveling, managing medications, and handling finances. The total score ranges from 0 to 8, with lower scores indicating a higher level of dependence.
Lawton Brody Activities of Daily Living Scale | 3 weeks
  The scale was developed in 1969 by Lawton and Brody to assess individuals' instrumental activities of daily living. This scale includes a total of eight items: using the telephone, shopping, preparing meals, housekeeping, doing laundry, traveling, managing medications, and handling finances. The total score ranges from 0 to 8, with lower scores indicating a higher level of dependence.
Lawton Brody Activities of Daily Living Scale | 6 weeks
  The scale was developed in 1969 by Lawton and Brody to assess individuals' instrumental activities of daily living. This scale includes a total of eight items: using the telephone, shopping, preparing meals, housekeeping, doing laundry, traveling, managing medications, and handling finances. The total score ranges from 0 to 8, with lower scores indicating a higher level of dependence.
Lawton Brody Activities of Daily Living Scale | 12 weeks
  The scale was developed in 1969 by Lawton and Brody to assess individuals' instrumental activities of daily living. This scale includes a total of eight items: using the telephone, shopping, preparing meals, housekeeping, doing laundry, traveling, managing medications, and handling finances. The total score ranges from 0 to 8, with lower scores indicating a higher level of dependence.

SECONDARY OUTCOMES:
Short Form 36 Quality of Life Scale | 1 day
  The SF-36 scale, developed by Ware in 1992, is commonly used for the assessment of quality of life. The SF-36 evaluates eight health dimensions: physical functioning, physical role, emotional role, pain, mental health, vitality, social functioning, and general health perception, comprising a total of 36 items. Item 2 assesses changes over the past year, while the remaining items focus on evaluations from the past four weeks. Items 4 and 5 are formatted in a yes/no response format, while the other items use Likert-type scales (3, 5, and 6-point). Additionally, questions numbered 1, 6, 7, 8, 9a, 9d, 9e, 9h, 11b, and 11d are reverse-coded, meaning their responses are inverted prior to score calculation. During the assessment, separate total scores are obtained for each subscale, and these scores range from 0 to 100. An increase in the SF-36 score indicates better quality of life, while a decrease signifies poorer quality of life.
Short Form 36 Quality of Life Scale | 2 day
  The SF-36 scale, developed by Ware in 1992, is commonly used for the assessment of quality of life. The SF-36 evaluates eight health dimensions: physical functioning, physical role, emotional role, pain, mental health, vitality, social functioning, and general health perception, comprising a total of 36 items. Item 2 assesses changes over the past year, while the remaining items focus on evaluations from the past four weeks. Items 4 and 5 are formatted in a yes/no response format, while the other items use Likert-type scales (3, 5, and 6-point). Additionally, questions numbered 1, 6, 7, 8, 9a, 9d, 9e, 9h, 11b, and 11d are reverse-coded, meaning their responses are inverted prior to score calculation. During the assessment, separate total scores are obtained for each subscale, and these scores range from 0 to 100. An increase in the SF-36 score indicates better quality of life, while a decrease signifies poorer quality of life.
Short Form 36 Quality of Life Scale | 3 weeks
  The SF-36 scale, developed by Ware in 1992, is commonly used for the assessment of quality of life. The SF-36 evaluates eight health dimensions: physical functioning, physical role, emotional role, pain, mental health, vitality, social functioning, and general health perception, comprising a total of 36 items. Item 2 assesses changes over the past year, while the remaining items focus on evaluations from the past four weeks. Items 4 and 5 are formatted in a yes/no response format, while the other items use Likert-type scales (3, 5, and 6-point). Additionally, questions numbered 1, 6, 7, 8, 9a, 9d, 9e, 9h, 11b, and 11d are reverse-coded, meaning their responses are inverted prior to score calculation. During the assessment, separate total scores are obtained for each subscale, and these scores range from 0 to 100. An increase in the SF-36 score indicates better quality of life, while a decrease signifies poorer quality of life.
Short Form 36 Quality of Life Scale | 6 weeks
  The SF-36 scale, developed by Ware in 1992, is commonly used for the assessment of quality of life. The SF-36 evaluates eight health dimensions: physical functioning, physical role, emotional role, pain, mental health, vitality, social functioning, and general health perception, comprising a total of 36 items. Item 2 assesses changes over the past year, while the remaining items focus on evaluations from the past four weeks. Items 4 and 5 are formatted in a yes/no response format, while the other items use Likert-type scales (3, 5, and 6-point). Additionally, questions numbered 1, 6, 7, 8, 9a, 9d, 9e, 9h, 11b, and 11d are reverse-coded, meaning their responses are inverted prior to score calculation. During the assessment, separate total scores are obtained for each subscale, and these scores range from 0 to 100. An increase in the SF-36 score indicates better quality of life, while a decrease signifies poorer quality of life.
Short Form 36 Quality of Life Scale | 12 weeks
  The SF-36 scale, developed by Ware in 1992, is commonly used for the assessment of quality of life. The SF-36 evaluates eight health dimensions: physical functioning, physical role, emotional role, pain, mental health, vitality, social functioning, and general health perception, comprising a total of 36 items. Item 2 assesses changes over the past year, while the remaining items focus on evaluations from the past four weeks. Items 4 and 5 are formatted in a yes/no response format, while the other items use Likert-type scales (3, 5, and 6-point). Additionally, questions numbered 1, 6, 7, 8, 9a, 9d, 9e, 9h, 11b, and 11d are reverse-coded, meaning their responses are inverted prior to score calculation. During the assessment, separate total scores are obtained for each subscale, and these scores range from 0 to 100. An increase in the SF-36 score indicates better quality of life, while a decrease signifies poorer quality of life.
Self-Care Agency Scale | 1 day
  The scale is used to assess an individual's ability to perform self-care. Developed by Kearney and Fleicher in 1979, it consists of 43 items. The scale evaluates four main characteristics of individuals: "active or passive response to situations," "motivation," "knowledge of health practices," and "self-esteem." The scale is answered using a 5-point Likert scale (0: Does not describe me at all, 1: Does not describe me well, 2: I am not sure, 3: Describes me somewhat, 4: Describes me very well). The lowest possible score on the scale is 35, and the highest score is 140. Higher scores indicate a greater ability and strength in self-care. There is no predetermined threshold or cut-off value for the Self-Care Scale.
Self-Care Agency Scale | 2 day
  The scale is used to assess an individual's ability to perform self-care. Developed by Kearney and Fleicher in 1979, it consists of 43 items. The scale evaluates four main characteristics of individuals: "active or passive response to situations," "motivation," "knowledge of health practices," and "self-esteem." The scale is answered using a 5-point Likert scale (0: Does not describe me at all, 1: Does not describe me well, 2: I am not sure, 3: Describes me somewhat, 4: Describes me very well). The lowest possible score on the scale is 35, and the highest score is 140. Higher scores indicate a greater ability and strength in self-care. There is no predetermined threshold or cut-off value for the Self-Care Scale.
Self-Care Agency Scale | 3 weeks
  The scale is used to assess an individual's ability to perform self-care. Developed by Kearney and Fleicher in 1979, it consists of 43 items. The scale evaluates four main characteristics of individuals: "active or passive response to situations," "motivation," "knowledge of health practices," and "self-esteem." The scale is answered using a 5-point Likert scale (0: Does not describe me at all, 1: Does not describe me well, 2: I am not sure, 3: Describes me somewhat, 4: Describes me very well). The lowest possible score on the scale is 35, and the highest score is 140. Higher scores indicate a greater ability and strength in self-care. There is no predetermined threshold or cut-off value for the Self-Care Scale.
Self-Care Agency Scale | 6 weeks
  The scale is used to assess an individual's ability to perform self-care. Developed by Kearney and Fleicher in 1979, it consists of 43 items. The scale evaluates four main characteristics of individuals: "active or passive response to situations," "motivation," "knowledge of health practices," and "self-esteem." The scale is answered using a 5-point Likert scale (0: Does not describe me at all, 1: Does not describe me well, 2: I am not sure, 3: Describes me somewhat, 4: Describes me very well). The lowest possible score on the scale is 35, and the highest score is 140. Higher scores indicate a greater ability and strength in self-care. There is no predetermined threshold or cut-off value for the Self-Care Scale.
Self-Care Agency Scale | 12 weeks
  The scale is used to assess an individual's ability to perform self-care. Developed by Kearney and Fleicher in 1979, it consists of 43 items. The scale evaluates four main characteristics of individuals: "active or passive response to situations," "motivation," "knowledge of health practices," and "self-esteem." The scale is answered using a 5-point Likert scale (0: Does not describe me at all, 1: Does not describe me well, 2: I am not sure, 3: Describes me somewhat, 4: Describes me very well). The lowest possible score on the scale is 35, and the highest score is 140. Higher scores indicate a greater ability and strength in self-care. There is no predetermined threshold or cut-off value for the Self-Care Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Turgut Şöhret, PhD student, Study Chair — Turgut ŞÖHRET
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] KATZ S, FORD AB, MOSKOWITZ RW, JACKSON BA, JAFFE MW. STUDIES OF ILLNESS IN THE AGED. THE INDEX OF ADL: A STANDARDIZED MEASURE OF BIOLOGICAL AND PSYCHOSOCIAL FUNCTION. JAMA. 1963 Sep 21;185:914-9. doi: 10.1001/jama.1963.03060120024016. No abstract available. PMID 14044222